CLINICAL TRIAL: NCT03198702
Title: Effectiveness and Safety of Early Intramuscular Botulinum Toxin Injections to Prevent Shoulder Deformity in Babies With Obstetrical Brachial Plexus Palsy
Acronym: POPB-TOX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POPB-TOX RB15.050
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Obstetrical Brachial Plexus Palsy
Keywords: physiotherapy; children; shoulder deformation; obstetrical brachial plexus palsy
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy | interventions — Botulinum Toxins, Type A; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: First group or "toxin" group: the babies will receive BOTOX injections at the age of 12 months in the shoulder muscles.
  Second group or "sham" group:the babies receive the same procedure but no injection.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toxin group (Experimental): The babies receive a botulinum toxin type A injection at the age of 12 months
  Interventions: Drug: Botulinum toxin type A injection
- Sham group (Sham Comparator): The babies receive a simulated injection procedure at the age of 12 months
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Botulinum toxin type A injection — A total of 8UI/kg will be injected in the internal shoulder rotator muscles: 2UI/kg in the sub scapular muscle, 3UI/kg in the pectoralis major muscle and 3UI/kg in the teres major/latissimus dorsi muscle.
  Arms: Toxin group
Other: Sham — The injection is mimed, the procedure is the same as the botulinum toxin injection.
  Arms: Sham group

SUMMARY:
In children population with obstetrical brachial plexus palsy (OBPP), shoulder musculoskeletal deformity is the main cause of morbidity, with a loss of range of shoulder motion, pain and a reduction in social participation. Some uncontrolled studies shows that early injections of botulinum toxin (BTI) in the internal shoulder rotator muscles (which cause the deformity) are one of the most promising treatment for the prevention of bony deformity.

The main objective of this study will be the evaluation of the effectiveness of BTI in the internal shoulder rotator muscles at the age of 12 months in preventing an increase in posterior subluxation of the glenohumeral joint in babies with OBPP (evaluated at the ages of 11 months and 18 months), compared to the Sham group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female babies with unilateral OBPP
* Age between 10 and 11 months
* Presenting one of 2 risk factors for posterior subluxation of the humeral head (10° less passive external ROM of the affected shoulder compared with the contralateral shoulder and/or a score strictly less than 6 on the AMS for shoulder external rotation and abduction, elbow flexion or supination)
* Signature of the consent form by (the) parent(s) over the age of majority

Exclusion Criteria:

* Bilateral OBPP
* Microsurgery or secondary muscle surgery planned between 12 and 18 months of age
* Contraindications to the use of botulinum toxin
* Contraindications to MRI
* MRI not possible in the Paediatric Day Hospital setting because of contraindications to the sedation protocol or due to organisational constraints
* Parents inapt to provide consent for the participation of their child
* Parents under the age of 18 years

Ages: 10 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage posterior migration of the humeral head measured on axial MRI slices between 11 (before the BTI carried out at 12 months) and 18 months of age (6 months post BTI). | At 18 month age

SECONDARY OUTCOMES:
compare the effectiveness of BTI with Sham procedure in preventing an increase in glenoid retroversion and three-dimensional deformity | At 18 month age
  With 2D glenoid changes measured on axial MRI and 3D glenoid version and migration of the humeral head measured on MRI
compare the effectiveness of BTI with Sham procedure in the improvement of active and passive joint range of motion and upper limb function | At 18 month age
  By measurement of passive range of motion, Active Movement Scale and Assistive Hand Assessment.
confirm good clinical tolerance of BTI treatment | At 18 month age
  By measurement of the number of serious and non-serious adverse events
evaluate the effects of BTI on trophicity, fibrosis and fatty infiltration of the injected muscles as well as muscle balance of the OBPP shoulder | At 18 month age
  Bu measurement of the degree of trophicity, fibrosis and fatty infiltration of the injected muscles (supraspinous, infraspinous, teres minor, subscapularis, teres major, pectoralis major, deltoid and latissimus dorsi)
determine if the treatment changes the frequency and type of surgical interventions in the long term | every years on 2 years old to 10 years old
  the number and type of surgical interventions undergone by the children in each group will be recorded during routine medical follow-up (as in usual practice) until the child's 10th birthday following unblinding (9 years and 6 months after the BTI).

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHRU Brest, Brest
  - Institut Régionnal de Réadaptation Centre de Réadaptation pour enfant, Flavigny-sur-Moselle
  - ESEAN (Etablissement de Santé pour Enfants et Adolescents de la région Nantaise), Nantes
  - CHU Nîmes, Nîmes
  - CHU Rennes, Rennes
  - CHU St Etienne, Saint-Etienne
  - Hôpital national de saint maurice, Saint-Maurice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pons C, Eddi D, Le Gal G, Garetier M, Ben Salem D, Houx L, Fitoussi F, Quintero N, Brochard S; POPB-TOX Group. Effectiveness and safety of early intramuscular botulinum toxin injections to prevent shoulder deformity in babies with brachial plexus birth injury (POPB-TOX), a randomised controlled trial: study protocol. BMJ Open. 2019 Sep 30;9(9):e032901. doi: 10.1136/bmjopen-2019-032901. PMID 31575585